CLINICAL TRIAL: NCT00961181
Title: Paclitaxel Releasing Balloon in Patients Presenting With In-Stent Restenosis A Prospective, Multi-centre, Non-randomized Clinical Trial With Follow-up Investigations at 1, 6 and 12 Months
Brief Title: Paclitaxel Releasing Balloon in Patients Presenting With In-Stent Restenosis
Acronym: PEPPER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Biotronik AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C0902
Record Dates: First submitted 2009-08-13; First posted 2009-08-18 (Estimated); Results first posted 2013-05-03 (Estimated); Last update posted 2013-05-06 (Estimated); Status verified 2013-05

CONDITIONS: In-stent Coronary Artery Restenosis
Keywords: paclitaxel; in-stent restenosis; BMS-ISR; DES-ISR; drug eluting balloon

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Paclitaxel Releasing Balloon (Experimental): Percutaneous coronary intervention with paclitaxel releasing balloon
  Interventions: Device: Paclitaxel Releasing Balloon

INTERVENTIONS:
Device: Paclitaxel Releasing Balloon — Percutaneous coronary intervention with paclitaxel releasing balloon
  Other Names: Pantera Lux

SUMMARY:
The primary objective of this study is to evaluate the safety and efficacy of the paclitaxel releasing balloon in patients with in-stent restenosis in a coronary artery.

DETAILED DESCRIPTION:
All patients are treated with the paclitaxel releasing balloon Pantera Lux. The indication is in-stent restenosis in either bare metal stent (BMS) or drug eluting stent (DES).

Clinical follow up visits at 1, 6 and 12 months. Angiographic follow up visit at 6 months.

ELIGIBILITY:
Inclusion Criteria:

1. Patient >/= 18 years
2. Written patient informed consent available
3. Patients with stable, unstable or documented silent angina pectoris
4. Patient eligible for percutaneous coronary intervention
5. Patient acceptable candidate for coronary artery bypass surgery
6. Patients with a single restenotic lesion in a previously stented area of a coronary artery (irrelevant whether BMS or DES related)
7. Target reference vessel diameter (visual estimation): 2 - 4 mm
8. Target lesion length (visual estimation): 8 - 28 mm
9. Target lesion stenosis (visual estimation): >/= 50% - < 100%

Exclusion Criteria:

1. Left ventricular ejection fraction of < 30%
2. Visible thrombus in the target vessel visualized by angiography
3. Myocardial infarction (STEMI/NSTEMI) within 72 hours of the intended treatment. Determination of CKMB and/or troponin T or I is required.

   Notes:

   Laboratory assessments to be done within 24 hours prior to intervention. Patients with CKMB and/or troponin T or I > 2 fold the upper limit of normal must not be included in the trial.
4. Patients with planned major surgery within 3 months after planned coronary intervention and/or risk of either acetylsalicylic acid of clopidogrel cessation
5. Lesion length longer than length of available treatment balloon
6. Impaired renal function (serum creatinine > 2.0mg/dl or 177 micro mol/l, determined within 72 hours prior to intervention)
7. Additional coronary lesions (restenotic or de novo) in the same vessel which requires treatment
8. Totally occluded coronary artery (Mehran classification IV and TIMI flow 0)
9. Target lesion located in vessel bifurcation
10. Previous and/or planned brachytherapy of target vessel
11. Target lesion located in left main coronary artery
12. Stroke or TIA < 6 months prior to procedure
13. Patient with signs of a cardiogenic shock
14. Patient under ongoing systemic immunosuppressive therapy with paclitaxel or agents of the -limus group (i.e. sirolimus, tacrolimus, everolimus)
15. Surgeries of any kind within 30 days prior to screening
16. Patient with bleeding diathesis in whom anticoagulation or antiplatelet medication is contraindicated
17. Known allergies to anti-platelet-, anticoagulation therapy, contrast media or paclitaxel
18. Pregnant and/or breast-feeding females or females who intend to become pregnant (pregnancy test required for females of child-bearing potential)
19. Patient with a life expectancy of less than one year
20. Patient currently enrolled in other investigational device or drug trial
21. Patient with known incompliance to medical (antiplatelet, anticoagulation) therapy
22. Patient not able or willing to adhere to follow-up visits including follow-up angiography

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2009-08; Primary Completion 2010-12 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Hehrlein, MD, Principal Investigator — University Medical Center, Freiburg i.Br., Germany
Locations (1):
- Prof. Dr. Christoph Hehrlein, Freiburg im Breisgau, Germany

REFERENCES:
- [Result] Hehrlein C, Dietz U, Kubica J, Jorgensen E, Hoffmann E, Naber C, Lesiak M, Schneider H, Wiemer M, Tolg R, Richardt G. Twelve-month results of a paclitaxel releasing balloon in patients presenting with in-stent restenosis First-in-Man (PEPPER) trial. Cardiovasc Revasc Med. 2012 Sep-Oct;13(5):260-4. doi: 10.1016/j.carrev.2012.06.002. Epub 2012 Aug 4. PMID 22867706

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From 14 August 2009 to 26 April 2010 a total of 81 patients at 9 heart centres in Europe were enrolled. Last follow-up was completed 09 May 2011.
Pre-assignment Details: No group assignment.
Groups:
- Paclitaxel Releasing Balloon: Patients meeting all inclusion and none of the exclusion criteria were enrolled and treated with the study device, the Pantera Lux paclitaxel releasing balloon, as per protocol.
Period: Overall Study
Arm/Group | Paclitaxel Releasing Balloon
Started | 81
Completed | 76
Not Completed | 5
Not completed — Death | 2
Not completed — Withdrawal by Subject | 2
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Groups:
- Paclitaxel Releasing Balloon: Patients meeting all inclusion and none of the exclsuion criteria were enrolled and treated with the study device, the Pantera Lux paclitaxel releasing balloon, as per protocol.
Arm/Group | Paclitaxel Releasing Balloon
Number analyzed (Participants) | 81
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 30
  >=65 years | 51
Age Continuous [Mean (Standard Deviation); unit: years] | 66 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 63
Region of Enrollment [Number; unit: participants]
  Germany | 67
  Poland | 9
  Denmark | 5

OUTCOME MEASURES:

1. Primary Outcome: In-stent Late Lumen Loss
Description: In-stent is defined as from proximal shoulder to distal shoulder of the dilated Pantera Lux balloon.
  Late lumen loss is defined as the difference between minimal luminal diameter after procedure and at 6 months, as evaluated by offline quantitative coronary angiography (QCA).
  Offline quantitative coronary angiography (QCA) analysis was performed by an independent core laboratory (Ulrich Dietz, MD, Deutsche Klinik für Diagnostik, Wiesbaden, Germany).
Time Frame: 6 months
Population: 2 patients died, 2 patients withdrew consent, 6 patients refused repeat angiography at 6 months follow up, 8 patients could not be analysed by QCA
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Paclitaxel Releasing Balloon
Number analyzed (Participants) | 63
mm | 0.07 (0.31)

2. Secondary Outcome: In-segment Late Lumen Loss
Description: In-segment is defined as from proximal shoulder to distal shoulder of the dilated Pantera Lux balloon plus 5 mm proximal and 5 mm distal.
  Late lumen loss is defined as the difference between minimal luminal diameter after procedure and at 6 months, as evaluated by offline quantitative coronary angiography (QCA).
  Offline quantitative coronary angiography (QCA) analysis was performed by an independent core laboratory (Ulrich Dietz, MD, Deutsche Klinik für Diagnostik, Wiesbaden, Germany).
Time Frame: 6 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Paclitaxel Releasing Balloon
Number analyzed (Participants) | 63
mm | 0.02 (0.32)

3. Secondary Outcome: Cumulative Major Adverse Cardiac Events Rate (Composite of Cardiac Death, Non-fatal Myocardial Infarction, Clinically Driven Target Lesion Revascularization, Clinically Driven Target Vessel Revascularization)
Description: All safety endpoint and serious adverse events were adjudicated by an independent clinical events committee.
  Major Adverse Cardiac Events = MACE Myocardial Infarction = MI Target Lesion Revascularization = TLR Target Vessel Revascularization = TVR
Time Frame: 6 months
Population: 2 patients died, 2 patients withdrew consent
Measure: Number; unit: participants
Arm/Group | Paclitaxel Releasing Balloon
Number analyzed (Participants) | 77
participants | 5

4. Secondary Outcome: Cumulative MACE Rate (Composite of Cardiac Death, Non-fatal MI, Clinically Driven TLR, Clinically Driven TVR)
Description: All safety endpoint and serious adverse events were adjudicated by an independent clinical events committee.
Time Frame: 12 months
Population: 2 patients died, 2 patients withdrew consent, 1 patient lost to follow up
Measure: Number; unit: participants
Arm/Group | Paclitaxel Releasing Balloon
Number analyzed (Participants) | 76
participants | 9

5. Secondary Outcome: In-stent Diameter Stenosis (%DS)
Description: In-stent is defined as from proximal shoulder to distal shoulder of the dilated Pantera Lux balloon.
  Diameter stenosis is defined as the difference between reference vessel diameter and minimal lumen diameter divided by reference vessel diameter x100%.
  Offline quantitative coronary angiography (QCA) analysis was performed by an independent core laboratory (Ulrich Dietz, MD, Deutsche Klinik für Diagnostik, Wiesbaden, Germany).
Time Frame: 6 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of re-narrowing
Arm/Group | Paclitaxel Releasing Balloon
Number analyzed (Participants) | 63
percentage of re-narrowing | 25.9 (11.7)

6. Secondary Outcome: In-segment Diameter Stenosis (%DS)
Description: In-segment is defined as from proximal shoulder to distal shoulder of the dilated Pantera Lux balloon plus 5 mm proximal and 5 mm distal.
  Diameter stenosis is defined as the difference between reference vessel diameter and minimal lumen diameter divided by reference vessel diameter x100%.
  Offline quantitative coronary angiography (QCA) analysis was performed by an independent core laboratory (Ulrich Dietz, MD, Deutsche Klinik für Diagnostik, Wiesbaden, Germany).
Time Frame: 6 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of re-narrowing
Arm/Group | Paclitaxel Releasing Balloon
Number analyzed (Participants) | 63
percentage of re-narrowing | 29.9 (10.6)

7. Secondary Outcome: Binary In-stent Restenosis
Description: In-sent is defined as from proximal shoulder to distal shoulder of the dilated Pantera Lux balloon.
  Binary restenosis was defined as a ≥ 50% diameter stenosis at follow-up as evaluated by offline quantitative coronary angiography (QCA).
  Diameter stenosis is defined as the difference between reference vessel diameter and minimal lumen diameter divided by reference vessel diameter x100%.
  Offline quantitative coronary angiography (QCA) analysis was performed by an independent core laboratory (Ulrich Dietz, MD, Deutsche Klinik für Diagnostik, Wiesbaden, Germany).
Time Frame: 6 months
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Paclitaxel Releasing Balloon
Number analyzed (Participants) | 63
participants | 2

8. Secondary Outcome: Binary In-segment Restenosis
Description: In-segment is defined as from proximal shoulder to distal shoulder of the dilated Pantera Lux balloon plus 5 mm proximal and 5 mm distal.
  Binary restenosis was defined as a ≥ 50% diameter stenosis at follow-up as evaluated by offline quantitative coronary angiography (QCA).
  Diameter stenosis is defined as the difference between reference vessel diameter and minimal lumen diameter divided by reference vessel diameter x100%.
  Offline quantitative coronary angiography (QCA) analysis was performed by an independent core laboratory (Ulrich Dietz, MD, Deutsche Klinik für Diagnostik, Wiesbaden, Germany).
Time Frame: 6 months
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Paclitaxel Releasing Balloon
Number analyzed (Participants) | 63
participants | 1

9. Secondary Outcome: Technical Success
Description: Technical success is defined as successful vascular access, completion of the endovascular procedure and immediate morphological success with < 30% residual diameter stenosis assessed by quantitative coronary angiography (QCA).
  Diameter stenosis is defined as the difference between reference vessel diameter and minimal lumen diameter divided by reference vessel diameter x100%.
  Offline quantitative coronary angiography (QCA) analysis was performed by an independent core laboratory (Ulrich Dietz, MD, Deutsche Klinik für Diagnostik, Wiesbaden, Germany).
Time Frame: directly after intervention (after finalized treatment)
Measure: Number; unit: participants
Arm/Group | Paclitaxel Releasing Balloon
Number analyzed (Participants) | 81
participants | 81

10. Secondary Outcome: Device Success
Description: Device success defined as exact deployment of the device as documented by two different projections assessed by quantitative coronary angiography (QCA).
  Offline quantitative coronary angiography (QCA) analysis was performed by an independent core laboratory (Ulrich Dietz, MD, Deutsche Klinik für Diagnostik, Wiesbaden, Germany).
Time Frame: directly after intervention (after finalized treatment)
Measure: Number; unit: participants
Arm/Group | Paclitaxel Releasing Balloon
Number analyzed (Participants) | 81
participants | 80

ADVERSE EVENTS:
Time Frame: 1 year
Description: On-site follow up at 6 and 12 month follow up. All safety endpoint and serious adverse events were adjudicated by an independent clinical events committee
Arm/Group | Paclitaxel Releasing Balloon
Serious Adverse Events (participants affected / at risk) | 11/76
Other Adverse Events (participants affected / at risk) | 0/76
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Paclitaxel Releasing Balloon (N=76)
Cardiac death (Cardiac disorders) | 0 (0)
Non-fatal myocardial infarction (Cardiac disorders) | 1 (1)
Target vessel revascularization (Vascular disorders) | 1 (1)
Target lesion revascularization (Vascular disorders) | 7 (7)
Non-cardiac death (General disorders) | 2 (2)
Stent thrombosis (Vascular disorders) | 0 (0)

LIMITATIONS AND CAVEATS:
Single arm design. Optimal time point for a quantitative angiographic follow up should be scheduled after 12 months, as recommended by the Academic Research Consortium guidelines for DES.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less